CLINICAL TRIAL: NCT02775045
Title: Eosinophil β1 Integrin Activation as a Biomarker for Eosinophilic Esophagitis
Acronym: EoE
Status: Completed | Type: Observational
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Other Study IDs: 2016-0508; R21AI122103-01A1 (NIH)
Record Dates: First submitted 2016-05-13; First posted 2016-05-17 (Estimated); Last update posted 2019-01-30 (Actual); Status verified 2019-01

CONDITIONS: Eosinophilic Esophagitis
Keywords: EoE
MeSH Terms: conditions — Eosinophilic Esophagitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 55 mL of blood will be drawn during V1 and V2. The blood will be drawn to save serum, for flow cytometry to answer the research questions, to isolate plasma and purify eosinophils for banking of whole cell protein and RNA, and to allow for genetic analysis of DNA. DNA will be isolated for directed genetic analysis of genes related to eosinophil biology and inflammation associated with EoE. Currently, these include ORMDL3, eotaxin-3, and IL-13 and may include others upon identification in the literature. This limited analysis is not expected to be sufficient for subject identification nor is it expected that the genes will be predictive of any other disease process. The genetic portion of the blood draw will not be optional.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Eosinophil esophagitis: Adult patients (>18 yr) will be recruited from the Gastroenterology clinic following a diagnostic endoscopy for esophageal dysfunction with predominant symptom(s) of solid food dysphagia and/or esophageal food impaction. Patients with esophageal biopsy showing greater than 15 eosinophil/hpf (pathology results typically available within three business days) despite greater than two months use of high dose proton pump inhibitor will be invited to participate and enroll in the study within 1 week of the endoscopy.
  Interventions: Other: Observation Period

INTERVENTIONS:
Other: Observation Period — 8 week observational period

SUMMARY:
The purpose of this study is to improve the overall management of patients with Eosinophil Esophagitis. Currently, the best way to monitor Eosinophil Esophagitis is repeating the endoscopy procedure. The investigators plan to identify a biomarker in the blood (a measurable substance) that tracks with disease activity and will reduce the need for follow-up endoscopies.

DETAILED DESCRIPTION:
By definition, Eosinophil Esophagitis involves the presence of eosinophils in the esophageal mucosa. Although incompletely understood, the pathophysiology of Eosinophil Esophagitis is thought to include food allergen driven inflammation in the esophageal mucosa that triggers release of mediators for recruitment of eosinophils. The mediators, such as eotaxin, invoke eosinophil activation and trafficking into the esophageal tissue. The subsequent release of mediators from eosinophils and other cells, including mast cells and basophils, promotes inflammation and fibrosis resulting in Eosinophil Esophagitis symptoms. This protocol focuses on early eosinophil activation events in Eosinophil Esophagitis in the peripheral circulation, specifically activation of surface β1 integrin, as a biomarker for disease activity reflecting eosinophils destined for trafficking into the esophagus. Demonstrating a correlation between disease activity and a peripheral biomarker may ultimately facilitate a timelier, less invasive and less costly management strategy for Eosinophil Esophagitis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female with no health concerns that might affect the outcome of the study,
* Age 18 years of age and older
* Esophageal dysfunction with a predominant symptom of solid food dysphagia and/or esophageal food impaction
* Esophageal eosinophilia (>15 eosinophils/HPF) shown on biopsy
* In the opinion of the investigator, capable and willing to grant written informed consent and cooperate with study procedures and requirements.

Exclusion Criteria:

* Major health problems such as autoimmune disease, heart disease, type I and II diabetes, uncontrolled hypertension or lung diseases other than asthma. The listed health problems are definitive exclusion but decisions regarding major health problems not listed will be based upon the judgment of the investigator,
* Pregnant or lactating females or has a planned pregnancy during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (>18 yr) will be recruited from the Gastroenterology clinic following a diagnostic endoscopy for esophageal dysfunction with predominant symptom(s) of solid food dysphagia and/or esophageal food impaction. Patients with esophageal biopsy showing greater than 15 EOS/hpf (pathology results typically available within three business days) despite greater than two months use of high dose proton pump inhibitor will be invited to participate and enroll in the study within 1 week of the endoscopy.
Sampling Method: Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2016-08-30 (Actual); Primary Completion 2018-12-13 (Actual); Study Completion 2018-12-13 (Actual)

PRIMARY OUTCOMES:
Eosinophil Esophagitis symptom score | 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Sameer Mathur, MD/PhD, Principal Investigator — UW Madison
Locations (1):
- UW Madison School of Medicine and Public Health, Madison, Wisconsin, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Derived] Bartig KA, Lee KE, Mosher DF, Mathur SK, Johansson MW. Platelet association with leukocytes in active eosinophilic esophagitis. PLoS One. 2021 Apr 23;16(4):e0250521. doi: 10.1371/journal.pone.0250521. eCollection 2021. PMID 33891621